CLINICAL TRIAL: NCT00763685
Title: Double-Blind, Randomized, Placebo -Controlled Study to Evaluate the Efficacy of Pre-operative Administration of Etoricoxib 120 mg, Etoricoxib 120 mg and Paracetamol 1 g Combination or Placebo in the Treatment of Postoperative Pain in Patients Undergoing Gynaecologic Laparoscopic Surgery
Brief Title: Study to Evaluate the Efficacy of Pre-operative Administration of Etoricoxib 120 mg, Etoricoxib 120 mg and Paracetamol 1 g Combination or Placebo in the Treatment of Postoperative Pain in Patients Undergoing Gynaecologic Laparoscopic Surgery
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The gynecological laparoscopic surgery transition to day surgery made following the study protocol not possible.
Sponsor: East Tallinn Central Hospital (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Tiina Arumagi, anaesthesiologist, East Tallinn Central Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 35195; EUDRACT 2008-004098-17
Record Dates: First submitted 2008-09-30; First posted 2008-10-01 (Estimated); Last update posted 2012-01-31 (Estimated); Status verified 2012-01

CONDITIONS: Pain
Keywords: preoperative pain prophylaxis; postoperative pain
MeSH Terms: conditions — Pain; Pain, Postoperative | interventions — Etoricoxib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- etoricoxib 120 mg (Active Comparator): active control
  Interventions: Drug: etoricoxib
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: etoricoxib
- 3 (Active Comparator): Paracetamol 1 g and etoricoxib 120 mg
  Interventions: Drug: etoricoxib

INTERVENTIONS:
Drug: etoricoxib — etoricoxib 120 mg, paracetamol 1 g

SUMMARY:
Primary Hypothesis:

1. The analgesic effect of etoricoxib 120 mg administered 1 hour preoperatively is greater than that of placebo in the treatment of postoperative pain.

ELIGIBILITY:
Inclusion Criteria:

1. Type of gynaecologic surgery:

   * diagnostic laparoscopy
   * sterilization
   * removal of ovarial cyst
   * chromopertubation
   * laparoscopic myomectomy
   * laparoscopic fenestration of ovaria
   * laparoscopic adhesiolysis
2. Age 18-50 years.
3. Evaluated risk of anaesthetic procedure according to ASA (American Society of Anaesthesiologist) classification: ASA I or II.
4. Patients agreed to participate in the study and signed the informed consent.

Exclusion Criteria:

1. ASA III or more
2. Emergency surgery
3. Major laparoscopic surgery i.e. hysterectomy
4. Duration of surgery more than 90 minutes
5. Chronic pain
6. History of hypersensitivity to the active substance or to any of the excipients of study drug (Paracetamol or Etoricoxib)
7. Active peptic ulceration or active gastro-intestinal (GI) bleeding.
8. Patients who have experienced bronchospasm, acute rhinitis, nasal polyps, angioneurotic oedema, urticaria, or allergic-type reactions after taking acetylsalicylic acid or NSAIDs including COX-2 (cyclooxygenase-2) inhibitors.
9. Pregnancy and lactation
10. Severe hepatic dysfunction (serum albumin < 25 g/l or Child-Pugh score ≥ 10).
11. Estimated renal creatinine clearance < 30 mL/min.
12. Children and adolescents under 16 years of age.
13. Inflammatory bowel disease.
14. Congestive heart failure (NYHA II-IV).
15. Patients with hypertension whose blood pressure has not been adequately controlled.
16. Established ischaemic heart disease, peripheral arterial disease, and/or cerebrovascular disease, unstable angina.
17. Patient has undergone coronary artery bypass graft surgery, angioplasty, or had myocardial infarction, cerebrovascular accident or transient ischemic attack within the past 6 months.
18. History of drug abuse.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2010-06; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Pain scale | 24 hours

SECONDARY OUTCOMES:
Vomiting | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Tiina Arumägi, MD, Principal Investigator — East Tallinn Central Hospital
Locations (1):
- East Tallinn Central Hospital, Tallinn, Estonia